CLINICAL TRIAL: NCT02856841
Title: The Preoperative Predictors of Optimal Cytoreductive Surgery in Women With Advanced Epithelial Ovarian Cancer
Brief Title: The Preoperative Predictors of Optimal Cytoreductive Surgery in Women With Advanced Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Other Study IDs: 152
Record Dates: First submitted 2016-08-01; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Ovarian Cancer
Keywords: epithelial ovarian cancer; optimum cytoreduction
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- optimum cytoreduction: without any gross tumor residue after surgery
- Suboptimum cytoreduction: with any gross tumor residue after surgery

SUMMARY:
44 patients were enrolled in this study as they had malignant epithelial ovarian tumor.Pre-operative staging was assessed by CT scan based on FIGO classification and compared to the standard laparotomy surgical staging. Maximal surgical effort for Optimum cytoreduction was achieved and the risk factors for sub-optimal cytoreduction were studied

DETAILED DESCRIPTION:
Each patient was subjected to comprehensive medical history taking and careful clinical examination, laboratory investigations (CA-125) and imaging (abdomino-pelvic CT scan). Patients with suspected bowel involvement were subjected for colonoscopy.

Pre-operative Abdomino-pelvic CT scans:

Preoperative CT scans were performed with a high-speed scanner after the oral and intravenous administration of contrast medium. The hard copy images were reviewed by consultant radiologists for assessment of the findings suggestive of malignant adnexal mass which are bilateral lesions, thick septa, enhancing solid components, ascites, and peritoneal deposits .

Pre-operative staging of cancer ovary was assessed by CT scan based on FIGO classification:

1. Stage II: tumor involving ovaries with pelvic extension +/- ascites.
2. Stage III: tumor involving ovaries with peritoneal implant outside pelvis +/- ascites.
3. Stage IV: tumor involving ovaries with parenchymal liver metastasis and/or pleural effusion.

Surgical treatment:

All patients underwent standard longitudinal laparotomy, intensive surgical staging and maximal surgical effort for Optimum cytoreduction which was included all of the following (total abdominal hysterectomy, bilateral salpingo-oophorectomy, infracolic-omentectomy, appendectomy, surgical removal of all tumor masses, intestinal resections if required).Achievement of no gross residual disease has been attempted in all cases. Finally, patients were divided into two groups:

* Suboptimal cytoreduction group with any gross tumor residue.
* Optimal cytoreduction group without any gross tumor residue.

Surgical risk factors for optimum cytoreduction:

* Parenchymal liver involvement.
* Omental involvement.
* Bowel involvement.
* Para aortic lymph node involvement.
* Peritoneal carcinomatosis: it is defined as disease > 4 mm involving 2 or more of the following areas; lateral colic gutters, anterior abdominal wall, diaphragm, and pelvic peritoneal reflections.
* Pelvic sidewall invasion: it is defined as presence of one or more of the following; tumor fixed to the pelvic bony wall, encasement of iliac vessels, and hydroureter.

ELIGIBILITY:
Inclusion Criteria:

* malignant epithelial ovarian tumor (EOC)

FIGO stage II, III, and IV.

Exclusion Criteria:

* Patients with previous abdominal or pelvic major surgery, synchronous abdominal or pelvic pathology or medically unfit for surgery

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 44 patients were enrolled in this study as they had malignant epithelial ovarian tumor (EOC), FIGO stage II, III, and IV.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
feasibility of optimum cytoreduction | 1 year after surgery
  ability to remove all gross lesions from the tumor intraoperatively and leaving no ovarian lesion seen by naked eye of the expert surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school

IPD SHARING:
Plan to Share IPD: Yes